CLINICAL TRIAL: NCT00827957
Title: A Phased Prospective Clinical Study Comparing Controlled Therapeutic Hypothermia Post Resuscitation After Cardiac Arrest Using External and Internal Cooling to Standard Intensive Care Unit Therapy
Brief Title: Comparing Therapeutic Hypothermia Using External and Internal Cooling for Post-Cardiac Arrest Patients
Acronym: Hypothermia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRB 2008/080/C
Record Dates: First submitted 2009-01-21; First posted 2009-01-23 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Cardiac Arrest
Keywords: Hypothermia; Internal cooling; External cooling; Cardiac arrest
MeSH Terms: conditions — Heart Arrest; Hypothermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- External Cooling (Active Comparator): The gel-coated external cooling device consists of four water circulating gel coated energy transfer pads, and is placed on the patient's back, abdomen, and both thighs. Depending on the size used, the total surface area ranges between 0.60 and 0.77 m2. It is connected to an automatic thermostat controlling the temperature of the circulating water (4°C to 42°C) based on the patient's core temperature.
  Interventions: Device: External Cooling
- Internal Cooling (Active Comparator): The intravascular cooling system uses a single lumen (8.5 Fr,38 cm) central venous catheter inserted into the inferior vena cava via the left or right femoral vein. Normal saline is pumped through three balloons mounted on the catheter and returned to a central system in a closed loop. The saline flow within the balloons is in close contact with the patient's blood flow and serves as a heat exchange system. An automatic temperature control device adjusts the temperature of the circulating saline (4°C to 42°C) based on the patient's core temperature.
  Interventions: Device: Internal Cooling

INTERVENTIONS:
Device: Internal Cooling — The intravascular cooling system uses a single lumen (8.5 Fr,38 cm) central venous catheter inserted into the inferior vena cava via the left or right femoral vein. Normal saline is pumped through three balloons mounted on the catheter and returned to a central system in a closed loop. The saline flow within the balloons is in close contact with the patient's blood flow and serves as a heat exchange system. An automatic temperature control device adjusts the temperature of the circulating saline (4°C to 42°C) based on the patient's core temperature.
  Other Names: Alsius Thermogard
  Arms: Internal Cooling
Device: External Cooling — The gel-coated external cooling device consists of four water circulating gel coated energy transfer pads, and is placed on the patient's back, abdomen, and both thighs. Depending on the size used, the total surface area ranges between 0.60 and 0.77 m2. It is connected to an automatic thermostat controlling the temperature of the circulating water (4°C to 42°C) based on the patient's core temperature.
  Other Names: Arctic Sun
  Arms: External Cooling

SUMMARY:
Controlled therapeutic hypothermia is a method of preserving neurological function post-resuscitation.It has been associated with improved functional recovery and reduced histological deficits in animal models of cardiac arrest.

DETAILED DESCRIPTION:
Three randomized clinical studies have been reported showing improved neurological outcome and reduced mortality in post-resuscitation patients treated with hypothermia compared to controls. Of the various methods of inducing hypothermia, internal cooling using an endovascular catheter and external cooling using gel pads with a water based circulating system have shown the most promise. There have not been any studies looking at outcomes between the two methods of cooling.

ELIGIBILITY:
Inclusion Criteria:

1. Sustained return of spontaneous circulation (ROSC) after cardiac arrest, for more than 30 min
2. Patients aged between 18 to 80 years.
3. Patients who are hemodynamically stable, with a systolic BP > 90 mmHg with or without inotropic support.
4. Patients comatose or unresponsive post-resuscitation

Exclusion Criteria:

1. Hypotension despite fluid and/or vasopressor support
2. Positive pregnancy test in women below 50 years
3. Premorbid status bedbound and uncommunicative

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Survival to hospital discharge | 30 days post arrest

SECONDARY OUTCOMES:
Neurological status of post-resuscitation patients | 1 year post discharge

CONTACTS AND LOCATIONS:
Overall Officials: Marcus EH Ong, MBBS, MPH, Principal Investigator — Singapore General Hospital
Locations (2):
- Singapore (2):
  - National Heart Centre Singapore, Singapore
  - Singapore General Hospital, Singapore

REFERENCES:
- [Derived] Ferreira Da Silva IR, Frontera JA. Targeted temperature management in survivors of cardiac arrest. Cardiol Clin. 2013 Nov;31(4):637-55, ix. doi: 10.1016/j.ccl.2013.07.010. PMID 24188226